CLINICAL TRIAL: NCT06594939
Title: Multicenter Phase II Study of Mosunetuzumab and Polatuzumab Vedotin With Split-Dose CHP Chemotherapy for Elderly Patients With Diffuse Large B-Cell Lymphoma
Brief Title: Mosunetuzumab and Polatuzumab Vedotin With Split-Dose CHP Chemotherapy for Elderly Patients With Diffuse Large B-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nirav Shah, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00056497
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: Mosunetuzumab; Polatuzumab vedotin
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Cyclophosphamide; Doxorubicin; Prednisone; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mosum-Pola-SD-CHP (Experimental): Each cycle is 28 days and consists of one "A" treatment on Day 1 and one "B" treatment on Day 15 for six cycles.
  Day 1 ("A" part of cycle) Polatuzumab Vedotin 1.8 mg/kg Intravenous (IV); Mosunetuzumab (Cycle 1A) 5 mg Subcutaneous (SC); Cyclophosphamide 375 mg/m^2 IV; Doxorubicin 25 mg/m^2 IV; Prednisone 50 mg Orally
  Day 2 ("A" part of cycle) Pegfilgrastim 6 mg SC
  Day 8 ("A" part of cycle) Mosunetuzumab 45 mg SC
  Day 15 ("B" part of cycle) Mosunetuzumab (Cycle 1B-6B) 45 mg SC; Cyclophosphamide 375 mg/m^2 IV; Doxorubicin 25 mg/m^2 IV; Prednisone 50 mg Orally
  Day 16 ("B" part of cycle) Pegfilgrastim 6 mg SC
  Interventions: Drug: Polatuzumab Vedotin; Drug: Mosunetuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Other: Pegfilgrastim

INTERVENTIONS:
Drug: Polatuzumab Vedotin — A combination of a monoclonal antibody and a chemotherapy drug.
  Other Names: Polivy
Drug: Mosunetuzumab — A monoclonal antibody.
  Other Names: Lunsumio
Drug: Cyclophosphamide — Chemotherapy drug, alkylating agent.
  Other Names: Cytoxan
Drug: Doxorubicin — Chemotherapy drug, anthracycline antibiotic.
  Other Names: Adriamycin
Drug: Prednisone — Steroid, anti-inflammatory
Other: Pegfilgrastim — Granulocyte stimulating factor, biologic response modifier.
  Other Names: filgrastim

SUMMARY:
This single-arm, interventional phase 2 study is designed to evaluate whether the inclusion of mosunetuzumab subcutaneous and polatuzumab vedotin (Mosun-Pola) to a split-dose CHP chemotherapy backbone will improve outcomes for elderly patients with a new diagnosis of diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This trial combines two novel agents, mosunetuzumab subcutatneous and polatuzumab vedotin (Mosun-Pola), with cytotoxic chemotherapy while allowing de-escalation in rapidly responding patients. After completing the first two cycles of Mosun-Pola-SD-CHP therapy, subjects will undergo an interim response assessment with positron emission tomography (PET) / computed tomography (CT) and minimal residual disease (MRD) testing (ClonoSEQ; Adaptive Biotechnology) prior to Cycle 3A. Patients who are interim PET-negative and MRD-negative will be placed on an abbreviated treatment regimen, where they will receive Mosun-Pola-SD-CHP therapy for only four cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 70-74 who are determined to be unfit or frail by the Cumulative Illness Rating Scale-Geriatric (CIRS-G) score with 5-8 comorbid conditions scored 2 or more than 1 comorbidity scored 3-4 are allowed.
2. Newly diagnosed, untreated, biopsy-proven CD20 positive diffuse large B-cell lymphoma (DLBCL) (including high-grade B-cell lymphoma and T-cell/histiocyte-rich large B-cell lymphoma). Patients with discordant bone marrow (i.e., involved by low-grade/indolent non-Hodgkin lymphoma) are eligible. Patients with transformed DLBCL from underlying low-grade disease are eligible. Patients with composite DLBCL and concurrent low-grade lymphoma are eligible. Patients with prior treatment for low-grade NHL with non-anthracycline based regimens are eligible.

   a. Short-course prednisone or equivalent steroid for symptom management is allowable for up to seven days.
3. Measurable disease by positron emission tomography (PET) / computed tomography (CT) using the Lugano criteria (lymph node >1.5 cm or extranodal site >1.0 cm).
4. Adequate biospecimen sample that meets current Adaptive Clonality ID Test specimen requirements for DLBCL.

   a. Note: the preferred ID specimen type is a formalin-fixed paraffin-embedded (FFPE) lymph node biopsy, either FFPE slides or scrolls, targeting 40 microns of material.
5. Left ventricular ejection fraction ≥50% by echocardiography or multigated acquisition (MUGA) scan.
6. Karnofsky Performance Score ≥50 or Eastern Cooperative Oncology Group (ECOG) scan 0-2.
7. Ann Arbor Stage II bulky, III, or IV disease.
8. Minimum life expectancy greater than 3 months (should be explicitly documented by the enrolling investigator).
9. Negative HIV test. Individuals with a positive HIV test at screening are eligible provided that, prior to enrollment, they are stable on antiretroviral therapy for at least 4 weeks, have a CD4 count ≥200/µL, and have an undetectable viral load, and have not had a history of opportunistic infection attributable to acquired immunodeficiency syndrome (AIDS) within the last 12 months.
10. For patients with hepatitis B virus antigen (HBsAg) or core antibody (HBcAb) seropositivity, patients must have a negative hepatitis B viral load and an appropriate prophylaxis plan must be in place during chemotherapy therapy treatment. For all patients that are hepatitis B core antibody positive, they should take entecavir prophylaxis (0.5 mg by mouth daily) until 1 year from completion of chemotherapy. Hepatitis B viral load should be checked on these patients prior to starting chemotherapy and every 3 months thereafter if initial hepatitis B viral load is negative (±1 week if chemotherapy cycle is delayed). If hepatitis B viral load is positive, hepatology or ID referral is recommended, and hepatitis B viral load should be checked monthly and every 3 months for 12 months after end of treatment.
11. For patients with hepatitis C Ab positivity, a viral load must be checked and negative for enrollment.
12. Negative SARS-CoV-2 antigen or polymerase chain reaction (PCR) test within 7 days prior to enrollment.
13. Had at least one dose of a COVID-19 vaccine approved or authorized for emergency use by the FDA.
14. Intrathecal chemotherapy for central nervous system prophylaxis can only be given at the discretion of the primary oncologist.

    a. Note: patients who received high-dose methotrexate are not eligible for the study.
15. For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agree to refrain from donating sperm, as defined below:

    1. With a female partner of childbearing potential or pregnant female partners, male participants must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for 6 months after the final dose of Mosun-Pola-SD-CHP. Male participants must refrain from donating sperm during this same period.
    2. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the Informed Consent Form.
16. Ability to understand a written informed consent document, and the willingness to sign it.
17. In the opinion of the enrolling investigator, subject must be deemed able to comply with the study intervention.

Exclusion Criteria:

1. Prior treatment for DLBCL with chemotherapy, immunotherapy, and biologic therapy.
2. Current Grade >1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease.
3. Prior allogeneic or autologous stem cell transplant.
4. Prior solid organ transplant.
5. Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).
6. Known or suspected chronic active Epstein-Barr Virus (EBV) infection.
7. History of progressive multifocal leukoencephalopathy (PML).
8. Current or within 6 months of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease.
9. Patients with SARS-CoV-2 antigen or PCR testing positivity within 30 days prior to Cycle 1 Day 1.

   a. Any patient with documented SARS-CoV-2 infection within 6 months prior to planned Cycle 1 Day 1 must have no persistent respiratory symptoms, no evidence of residual sequelae, and have a negative PCR test for SARS-CoV-2.
10. Administration of a live, attenuated vaccine within 4 weeks before start of study therapy or anticipation that such a live, attenuated vaccine will be required during the study.
11. On immunosuppressant therapy for an active autoimmune disease, including, but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    a. Exceptions may be made for patients with a remote history of or well-controlled autoimmune disease, excluding patients on systemic immunosuppression for autoimmune disease, or patients who received such immunosuppression within 1 year prior.
12. Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
13. Recent major surgery within 4 weeks before the start of C1D1 with the exception of lymph node biopsies for diagnosis.
14. Prior treatment with radiotherapy within 2 weeks prior to Cycle 1 Day 1.

    1. If patients have received radiotherapy within 4 weeks prior to the initiation of study treatment, patients must have at least one measurable lesion outside of the radiation field to be eligible.
    2. Patients who have only one measurable lesion that was previously irradiated but subsequently progressed are eligible.
15. History of previous anthracycline exposure.
16. CNS or meningeal involvement at diagnosis.
17. Richter's Transformation (e.g., DLBCL transformed from an underlying chronic lymphocytic leukemia (CLL) ).
18. Patients with primary mediastinal large B cell lymphoma (PMBCL).
19. Creatinine clearance <40 mL/min by Cockcroft-Gault.
20. Poor hepatic function, defined as total bilirubin concentration greater than 3.0 mg/dL or transaminases over 4 times the maximum normal concentration, unless these abnormalities are felt to be related to the lymphoma (which should be explicitly documented by the enrolling physician).
21. Pulmonary dysfunction, defined as receiving supplemental O2 or significant pulmonary comorbidities (e.g., history of pneumonitis, severe chronic obstructive pulmonary disease (COPD) ).
22. Significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, congestive heart failure, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease.
23. Active infectious disease (if patient is on medications for such situations, enrolling physician should explicitly document justification of meeting this criteria).
24. Known concurrent bone marrow malignancies (e.g., myelodysplastic syndrome) or poor bone-marrow reserve, defined as neutrophil count less than 1.5 × 10^9/L or platelet count less than 100 × 10^9/L, unless caused by bone-marrow infiltration with lymphoma.
25. History of a second concurrent active malignancy or prior malignancy which required chemotherapy treatment within the preceding 2 years (other than cured basal or squamous cell carcinoma, low-risk prostate cancer on observation, and other in situ carcinomas that were completely treated).
26. Treatment with any investigational drug within 30 days before enrollment.
27. Unable or unwilling to sign consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response | Up to six months.
  This is defined as the number of subjects achieving a complete response at the end of treatment using the Lugano criteria.

SECONDARY OUTCOMES:
Partial Response | Up to six months
  This is defined as the number of subjects achieving a partial response at the end of treatment using the Lugano criteria.
Duration of Response | Up to 60 months
  This is defined as the time from the first documentation of tumor response to disease progression (per the Lugano criteria), relapse, or death among patients who achieve a response of partial response or better. The measure will be the median duration of response in months.
Overall Survival | 2 years
  This outcome measure is the number of subjects expiring from any cause.
Adverse Events | Up to 7 months
  The number of grade 3 or higher adverse events possibly, probably, or definitely related to study therapy in the safety run-in population from the start of therapy through 30 days after the end of study therapy. Adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, version 5.0. Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded using the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading system described by Lee et al., 2019. The scale for ICANS will be the ASTCT ICANS consensus grading for adults. The score evaluates neurotoxicity domains. The lowest grade is 1 (less severe) and the highest is 4 (more severe). The ASTCT Consensus Grading for CRS, is based on the severity of the patient's symptoms. The lowest grade is 1 and the highest is 4. The higher the grade, the more severe.
Study therapy completion | Up to 6 months
  The number of subjects who complete the study therapy.
Eligibility for abbreviated therapy | 56 days
  The number of subjects eligible for abbreviated therapy.
Eligibility for full therapy | 56 days
  The number of subjects eligible for full therapy.
CRS or ICANS | 28 days
  The number of subjects experiencing a CRS or ICANS of the total study population within the first 28 days after study therapy start. The scale for ICANS will be the ASTCT ICANS consensus grading for adults. The score evaluates various neurotoxicity domains. The lowest grade is 1 and the highest is 4. The higher the grade, the more severe the symptoms. The scale for CRS, ASTCT Consensus Grading for CRS, is based on the severity of the patient's symptoms. The lowest grade is 1 and the highest is 4. The higher the grade, the more severe the symptoms.
Minimal residual disease at Cycle 3 | 56 days
  The number of subjects who achieve minimal residual disease negativity at Cycle 3. This will be determined using the clonoSEQ assay.
Minimal residual disease at end of study treatment | Up to six monts
  The number of subjects who achieve minimal residual disease negativity at the end of treatment. This will be determined using the clonoSEQ assay.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, MD, Study Chair — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No